CLINICAL TRIAL: NCT06727123
Title: The Effect of Motivational Interviewing on Diabetes Self-Management in Type 2 Diabetic Patients
Brief Title: The Effect of Motivational Interviewing on Diabetes Self-Management in Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Sule Calisir Kundakci, Lecturer, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SCK22T24
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Motivational interviews will be conducted with diabetic patients for 6 months. Patients will be trained before starting the interviews.
  Interventions: Other: motivational interviewing
- Control (Experimental): No application will be made. Routine follow-ups will be made.
  Interventions: Other: Control

INTERVENTIONS:
Other: motivational interviewing — Motivational interviews will be conducted with diabetic patients for 6 months. Patients will be trained before starting the interviews.
  Arms: Motivational Interviewing
Other: Control — No application will be made. Routine follow-ups will be made.
  Arms: Control

SUMMARY:
Diabetes is a chronic metabolic disorder characterized by high blood sugar due to problems with insulin production or function. Its prevalence has increased significantly in recent decades due to sedentary lifestyles, unhealthy diets, and increasing obesity rates. Type 2 diabetes, in particular, is a major global and national health problem with projections showing that it continues to grow. Effective diabetes management requires patients to adopt healthy behaviors such as following a diet plan, monitoring blood sugar, increasing physical activity, and avoiding risky habits such as smoking. Inadequate adherence to treatment can lead to serious complications such as cardiovascular disease and kidney damage, which can be a burden to patients, families, and healthcare systems. Motivational interviewing, a patient-centered approach, helps individuals overcome resistance to behavioral change. This study was designed experimentally to determine the effect of motivational interviewing on diabetes self-management in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes is defined as a chronic metabolic disorder characterized by high blood sugar levels. Abnormalities in insulin production, function, or both are considered the primary causes of the disease. The epidemiology of diabetes has changed significantly over the last three decades. Diabetes mellitus is one of the most important health problems for both patients and society due to its high mortality, morbidity, and associated costs. The prevalence of diabetes continues to increase globally, driven by advances in technology, sedentary lifestyles, and increasing rates of obesity. Among these factors, the shift towards less active lifestyles plays a central role, with many individuals spending long periods sitting or engaging in low-energy activities. In addition, poor dietary habits, including increased consumption of high-calorie, processed foods, have increased the risk of developing diabetes, especially type 2 diabetes. In Turkey, the prevalence of type 2 diabetes reported in 2020 has shown a significant increase and is expected to increase further by 2050 if current trends continue. Effective treatment for diabetes requires patients to adopt positive attitudes and behaviors towards managing their health. However, many individuals have difficulty maintaining long-term lifestyle changes. Poor adherence to treatment plans and poor disease management often lead to a variety of complications, including acute and chronic health problems. These complications, such as cardiovascular disease, neuropathy, and kidney damage, impose a significant caregiving burden on individuals with diabetes, their families, and society as a whole. To alleviate these problems, individuals must engage in effective self-management to control their disease and prevent complications. Self-management refers to the individual's responsibility to maintain and improve their health. Diabetes self-management aims to normalize blood sugar levels and reduce the risk of long-term complications. Key practices include developing a personalized nutrition plan, monitoring blood sugar levels, maintaining metabolic control, increasing physical activity, and avoiding risky behaviors such as smoking or excessive alcohol consumption. Despite its importance, individuals living with diabetes often face challenges in adopting the lifestyle, behavioral, and psychological changes necessary for effective management. Motivational interviewing is an evidence-based approach that helps individuals resolve the dilemma of behavioral change and facilitates treatment adherence for chronic conditions such as diabetes. This patient-centered method emphasizes understanding the patient's unique challenges and goals, tailoring strategies to their specific needs, and encouraging autonomy. This study aims to evaluate the impact of motivational interviewing on diabetes self-management in patients with type 2 diabetes. It seeks to understand whether this approach can improve health outcomes by encouraging better adherence to treatment plans and supporting sustainable behavioral change, ultimately enhancing disease management in individuals coping with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who agree to participate in the study voluntarily, can speak and understand Turkish, can communicate comfortably, have no hearing, comprehension or vision problems, are literate, use a smartphone, have Type 2 Diabetes and have HbA1c ≥ 7% will be included in the study.

Exclusion Criteria:

* Patients with cognitive dysfunction and those using antipsychotic medication will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Diabetes Self-Management | 6 months
  Type 2 Diabetes Self-Management Scale

SECONDARY OUTCOMES:
HbA1c | 6 months
  Routine blood value monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR